CLINICAL TRIAL: NCT02102074
Title: Intra-peritoneal Environmental Changes Following Colorectal Surgery for Cancer
Brief Title: Intra-peritoneal Environmental Changes Following Surgery
Acronym: CRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0036
Record Dates: First submitted 2013-02-07; First posted 2014-04-02 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2013-02

CONDITIONS: Tumor Cells and Tumor Markers in Peritoneal Cavity
Keywords: colon and rectal tumors; colon cancer markers
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fluids from abdomen drain system
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators hypothesize that the presence of tumor cells and tumor markers in peritoneal cavity are indicative for peritoneal spread during surgery, and may serve as early markers for systemic and/or intra-peritoneal recurrence of the disease and ultimately improve our understanding of tumor spread and disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* colon and rectal cancer

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colon and rectal cancer patients
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
tumor cells and tumor markers | 2 years

SECONDARY OUTCOMES:
Cytokine levels in the abdomen | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Avital, M.D., Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba, Israel
  - Meir medical center, Kfar Saba, Israel